CLINICAL TRIAL: NCT05920642
Title: Risk-benefit Analysis of Intrathecal Morphine Administration to Patients Undergoing Surgical Treatment of Proximal Femoral Fracture (Monocentric, Single-blinded, Randomized Clinical Study Compared to Standard Treatment)
Brief Title: Postoperative Pain Relieve for Patients Undergoing Surgical Treatment of Femoral Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNO-KARIM2021-1; 2021-002765-17 (EudraCT Number)
Record Dates: First submitted 2023-06-07; First posted 2023-06-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Proximal Femur Fracture
Keywords: proximal femur fracture; morphine administration; pain relief; intrathecal administration; parenteral administration; surgery
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into two parallel groups.
Who Masked: Participant
Masking Description: The participant will not know which arm of the study he/she has been enrolled into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine administration (Experimental): Study subjects randomized into this arm will be administered morphine intrathecally in the dose of dose 100 ug.
  Interventions: Drug: Intrathecal morphine administration
- Parenteral administration of analgesics (Active Comparator): Study subjects randomized into this arm will receive standard postoperative pain management (parenteral administration of analgesics).
  Interventions: Drug: Parenteral administration of analgesics

INTERVENTIONS:
Drug: Intrathecal morphine administration — Administration of morphine into the spinal canal.
  Arms: Intrathecal morphine administration
Drug: Parenteral administration of analgesics — Standard postoperative pain management of analgesics using parenteral route of administration.
  Arms: Parenteral administration of analgesics

SUMMARY:
The aim of the study is to investigate postoperative pain relief for patients undergoing surgical treatment of proximal femoral fracture using intrathecal administration of morphine.

DETAILED DESCRIPTION:
In this study, the investigators will compare the efficiency of intrathecal morphine administration with the standard of care (parenteral application of analgesics) for pain relief in patients after proximal femoral fracture surgery. The secondary outcome measure will be to determine the frequency of adverse effects of intrathecally administered morphine. The study will be monocentric, randomized, and single-blinded. A total of 50 patients are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* 60 to 90 years of age
* surgical treatment of proximal femur fracture
* The American Society of Anesthesiologists (ASA) classification I to III
* spinal anesthesia used for the operation

Exclusion Criteria:

* general anesthesia used for the operation
* allergy to opioids
* high risk of respiratory depression

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Every 2 hours after the surgery, total of 24 hours
  Pain intensity will be assessed using the Visual Analogue Scale (VAS10) scale (0-10). The total value of all measured values will be calculated. The maximum value observed during the 24 hours will be also recorded.
Pain assessment during patient positioning | 24 hours
  Pain intensity will be assessed using the VAS10 scale (0-10) during the positioning of the patient.
Time to administration of rescue medication | 24 hours
  The time to administration of rescue medication (analgesics) will be observed in hours.
Total consumption of opioids on Intensive Care Unit | 24 hours
  The total consumption of opioids on Intensive Care Unit will be measured in the number of administered doses.

SECONDARY OUTCOMES:
Hypoventilation - bradypnea | 24 hours
  The observed parameters of hypoventilation include bradypnea = respiratory rate (RR)<10/min
Hypoventilation - presence of hypopnea (TV < 4) | 24 hours
  The observed parameters of hypoventilation will include hypopnea = Tidal Volume (TV) < 4 ml/min. It is a physiological parameter that fluctuates depending on the load in the range of 6-180 liters/min.
Hypoventilation - SpO2 | 24 hours
  The observed parameters of hypoventilation will include inability to maintain oxygen saturation (SpO2) above 90 % without the need for oxygenotherapy.
Hypoventilation - presence of hypoxemia (paO2) (below 10 kPa) | 24 hours
  The observed parameters of hypoventilation will include hypoxemia according to the analysis of blood gasses. Hypoxemia is diagnosed when the partial pressure of oxygen in the arterial blood (paO2) falls below 10 kiloPascals (kPa).
Hypoventilation - other signs of respiratory insufficiency | 24 hours
  The observed parameters of hypoventilation will include other signs of respiratory insufficiency. Will be evaluated as 0-no, 1-yes + the need for oxygenotherapy, 2-yes+ the need for antidote or other treatment
Hypotension | 24 hours
  The observed parameters of hypotension will be as follows: systolic blood pressure (SBP) < 90 mmHg and/or mean arterial pressure (MAP) < 60 mmHg and/or decrease of blood pressure (BP) by more than 20-30 % of the initial values. Evaluation: 0-no, 1-yes, without administration of noradrenaline, 2-yes, with noradrenaline administration.
Bradycardia | 24 hours
  The observed parameters of bradycardia will be as follows: heart rate (HR) < 50/min. Evaluation: 0-no, 1-yes + administration of atropine or ephedrine, 2-yes+ administration of atropine repeatedly or other treatment.
Postoperative nausea and vomiting | 24 hours
  The incidence of postoperative and vomiting will be observed. Evaluation: 0-no, 1-nausea, 2-vomiting
Effect of antiemetics | 24 hours
  The effect of antiemetics will be observed. Evaluation: 0-not administered, 1-administered, 2-no effect
Pruritus | 24 hours
  The presence and condition of pruritus will be observed. Evaluation: 0-no, 1-yes, no scratching, 2-moderate, need of scratching, 3-strong, need of treatment.
Effect of pruritus treatment | 24 hours
  The effect of pruritus treatment will be observed. Evaluation: 0-no medication administered, 1-administered, 2-no effect

CONTACTS AND LOCATIONS:
Overall Officials: Denis Buršík, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the individual participant data public.

REFERENCES:
- [Background] Rathmell JP, Pino CA, Taylor R, Patrin T, Viani BA. Intrathecal morphine for postoperative analgesia: a randomized, controlled, dose-ranging study after hip and knee arthroplasty. Anesth Analg. 2003 Nov;97(5):1452-1457. doi: 10.1213/01.ANE.0000083374.44039.9E. PMID 14570664
- [Background] Yamashita K, Fukusaki M, Ando Y, Tanabe T, Terao Y, Sumikawa K. Postoperative analgesia with minidose intrathecal morphine for bipolar hip prosthesis in extremely elderly patients. J Anesth. 2009;23(4):504-7. doi: 10.1007/s00540-009-0817-5. Epub 2009 Nov 18. PMID 19921358
- [Background] Kwan AS, Lee BB, Brake T. Intrathecal morphine for post-operative analgesia in patients with fractured hips. Hong Kong Med J. 1997 Sep;3(3):250-255. PMID 11847368